CLINICAL TRIAL: NCT01089504
Title: Prophylactic Phenobarbital After Resolution of Neonatal Seizures
Brief Title: Prophylactic Phenobarbital After Neonatal Seizures
Acronym: PROPHENO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate rate of enrollment
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ronnie Guillet, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 28907
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Neonatal Seizures
Keywords: phenobarbital; neonate; antiepileptic drugs; neurodevelopmental outcome; seizure
MeSH Terms: conditions — Seizures | interventions — Phenobarbital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenobarbital (Active Comparator): Phenobarbital, 4-5 mg/kg/day, for 4 months
  Interventions: Drug: phenobarbital
- Placebo (Placebo Comparator): Placebo in a volume equivalent to active drug for 4 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: phenobarbital — Phenobarbital, 4-5 mg/kg/d, by mouth, for 4 months
  Arms: Phenobarbital
Drug: placebo — Matched placebo, same volume as active drug, by mouth daily for 4 months
  Arms: Placebo

SUMMARY:
The treatment of infants with medications after their seizures have stopped is very variable. No one knows if continuing treatment with phenobarbital for up to several months is helpful or harmful. This clinical trial is designed to help answer that question and provide data that will help determine standard of care for these children.

DETAILED DESCRIPTION:
The treatment of infants with antiepileptic medications after the resolution of neonatal seizures is highly variable and controversial. Infants are commonly treated with phenobarbital after their seizures have resolved to prevent recurrence. Data to support this practice are lacking but animal models suggest that the neonatal brain is vulnerable to repeated seizures. Yet exposure of the developing brain to phenobarbital for prolonged periods may have deleterious consequences. We are proposing a multi-center, randomized, clinical trial (RCT) to determine if continued treatment with phenobarbital reduces seizure recurrence without adversely affecting neurodevelopmental outcome or if infants' outcomes are improved if no prophylactic medication is given. We will identify infants with seizures beginning in the first week that resolve within 7 days and randomize them to receive phenobarbital or placebo daily for four months. Via visits and frequent telephone contacts over the first six months, we will determine the rate of seizure recurrence. The primary outcome, neurodevelopmental status, will be assessed at 18-22 months using the Bayley Scales of Infant Development. Additional subgroup analyses are planned to determine the contribution of seizure etiology to outcome and predictive value of initial EEG classification. The trial will be conducted at 18 - 20 sites, chosen for their experience and proven track record for enrollment and retention in this specific population. The trial will be coordinated by the Clinical Trials Coordination Center at the University of Rochester and overseen by a Steering Committee composed of experienced trialists representing neonatology and pediatric neurology, biostatistics, and clinical trial administration.

Extrapolation from the results of an RCT of phenobarbital prophylaxis after febrile seizures in children suggests that phenobarbital may adversely affect brain development and may be ineffective in preventing seizures. Based on this previous RCT that resulted in near universal change in practice (the elimination of prolonged use of phenobarbital after simple febrile seizures), we anticipate that the data we generate may have a similar impact on standard of care for infants with neonatal seizures.

ELIGIBILITY:
Inclusion Criteria:

* Birth at > 34 weeks' gestation
* Neonatal seizures (clinical, electrographic or both), with onset in the first 120 hours after birth and resolution within 7 days of onset
* Parental informed consent

Exclusion Criteria:

* Birth at < 34 weeks' gestation
* If the attending neonatologist attributes the seizures solely to a transient abnormality, easily correctable and unlikely to recur (eg, transient electrolyte abnormalities). If the attending neonatologist cannot be contacted, the site PI will be asked to review the available information and judge whether the infant is eligible.
* If the infant has been diagnosed with or there is a strong suspicion of an inborn error of metabolism, significant brain malformation, microcephaly (< 3 %ile), or a chromosomal abnormality which, in the absence of seizures, is known to be independently associated with an increased likelihood of cognitive impairment
* If the infant has been diagnosed with an intrauterine viral infection
* If the infant is not expected to survive to discharge

Ages: 2 Days to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Guillet, MD, PhD, Principal Investigator — University of Rochester
Locations (18):
- United States (18):
  - University of Arkansas, Little Rock, Arkansas
  - University of California San Francisco, San Francisco, California
  - Univeristy of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Women & Children's Hospital of Buffalo, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenobarbital | Placebo
Started | 8 | 5
Completed | 5 | 4
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenobarbital | Placebo | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 5 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Bayley Scales of Infant Development (BSID) Score - Cognitive
Description: The Bayley Scales of Infant Development (BSID) measure the mental and motor development and test the behavior of infants from one to 42 months of age. The test is intended to measure a child's level of development in three domains: cognitive, motor, and behavioral. The primary outcome is the Bayley assessment of development at 2 years of age. This is a standardized developmental exam that is normalized to the age of the child in months. The mean adjusted score is 100 with a standard deviation of 15 (higher being better) - very similar to the more familiar IQ score.
Time Frame: 18-22 months
Population: Due to low enrollment, there was limited data available for analysis and therefore insufficient power to provide meaningful results for our primary or secondary analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenobarbital | Placebo
Number analyzed (Participants) | 8 | 5
units on a scale | 87.50 (11.90) | 92.50 (26.61)

2. Secondary Outcome: Mean Bayley Scales of Infant Development (BSID) Score - Motor
Description: This part of the BSID assesses the degree of body control, large muscle coordination, finer manipulatory skills of the hands and fingers, dynamic movement, postural imitation, and the ability to recognize objects by sense of touch.
Time Frame: 18-22 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phenobarbital | Placebo
Number analyzed (Participants) | 8 | 5
units on a scale | 82.80 (24.59) | 83.75 (20.65)

3. Secondary Outcome: Number of Participants With One or More Seizures
Description: Any clinical or electrographic seizures occurring between study entry and all follow-up examinations and contacts.
Time Frame: 18-22 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Phenobarbital | Placebo
Number analyzed (Participants) | 8 | 5
participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | Phenobarbital | Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/5
Other Adverse Events (participants affected / at risk) | 6/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phenobarbital (N=8) | Placebo (N=5)
failure to thrive (Metabolism and nutrition disorders) | 0 | 1
poor quality sleep (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phenobarbital (N=8) | Placebo (N=5)
apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
convulsion (Nervous system disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 1 — fever
upper respiratory tract infection (Infections and infestations) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 — blood in stool
seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
flatulence (Gastrointestinal disorders) | 0 | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 0
status epilepticus (Nervous system disorders) | 1 | 0
poor quality sleep (Nervous system disorders) | 1 | 0
influenza (Infections and infestations) | 1 | 0
ear infection (Ear and labyrinth disorders) | 2 | 0
gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
sinusitis (Infections and infestations) | 1 | 0
otitis media (Ear and labyrinth disorders) | 4 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
Croup infection (Infections and infestations) | 1 | 0
Candidiasis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus infection (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to low enrollment, there was limited data available for analysis and therefore insufficient power to provide meaningful results for our primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes